CLINICAL TRIAL: NCT05794919
Title: Bioequivalence Study of Calcium Hydroxybenzene Sulphonate Dispersible Tablets and Calcium Hydroxybenzene Sulfonate Tablets (Doxium®) Under Fed Conditions in Chinese Healthy Volunteers
Brief Title: Bioequivalence Study of Calcium Hydroxybenzene Sulphonate Dispersible Tablets in Chinese Healthy Volunteers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tongren Hospital (Other)
Collaborators: Hainan Linheng Pharmaceutical Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2022-BE-QBHSGFSP-04
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Bioequivalence Study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calcium Hydroxybenzene Sulphonate Dispersible Tablets (Experimental): The healthy subjects will be administered a single dose of Calcium Hydroxybenzene Sulphonate Dispersible Tablets 0.25g under fast or fed conditions.
  Interventions: Drug: Calcium Hydroxybenzene Sulphonate Dispersible Tablets 0.25g
- Doxium® (Active Comparator): The healthy subjects will be administered a single dose of Doxium® 250mg under fast or fed conditions.
  Interventions: Drug: Calcium Hydroxybenzene Sulfonate Tablets（Doxium®) 250mg

INTERVENTIONS:
Drug: Calcium Hydroxybenzene Sulphonate Dispersible Tablets 0.25g — A generic product manufactured by Hainan Linheng Pharmaceutical Co., Ltd.
  Arms: Calcium Hydroxybenzene Sulphonate Dispersible Tablets
Drug: Calcium Hydroxybenzene Sulfonate Tablets（Doxium®) 250mg — Calcium Hydroxybenzene Sulfonate Tablets（Doxium®）produced by OM pharma S.A.
  Arms: Doxium®

SUMMARY:
The aim of this study is to evaluate the bioequivalence of two Calcium Hydroxybenzene Dispersible Tablets in healthy Chinese volunteers.

DETAILED DESCRIPTION:
The trial preparation is Calcium Hydroxybenzene Sulphonate Dispersible Tablets produced by Hainan Linheng Pharmaceutical Co., Ltd.

The reference preparation is Calcium Hydroxybenzene Sulphonate Tablets (Doxium ®) produced by OM pharma S.A.

The bioequivalence of two preparations will be evaluated at the fast or fed conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Participate voluntarily and sign an informed consent form before the study;
2. Age: 18 to 55 years old (including 18 and 55 years old) , male and female;
3. Weight: female subjects with weight ≥45.0kg, male subjects with weight ≥50.0kg, with the body mass index of 19.0~28.0 kg/m (including 19.0 and 28.0);
4. The physical examination, vital signs, laboratory examination and electrocardiogram are not abnormal or abnormal but with no clinical significance;
5. Have no pregnancy plan and appropriate contraceptive measures during the trial and within 6 months after the last dose.
6. Be able to communicate well, understand and comply with the requirements of the study.

Exclusion Criteria:

1. Be allergic, or have a clear history of allergies to trial drugs and excipients;
2. Have diseases in circulatory system, respiratory system, digestive system, hematologic system, nervous system, immune system, urinary system, endocrine system and mental system, or have medical history of the above-mentioned systems and other diseases that may significantly affect drug absorption, distribution, metabolism and excretion.
3. Have a history of drug abuse or are positive for urine durg screening;
4. Pregnant or lactating women, or serum HCG positive for female subjects, or there was a unprotected sex within 2 weeks before screening;
5. Frequent smokers and alcoholics within the first 3 months (smoking more than 5 cigarettes/day on average, drinking an average of more than 21 units of alcohol per week, 1 unit = 360 mL beer or 45 mL liquor or 150 mL wine), or cannot stop using any tobacco products, or unable to stop alcohol intake during the whole research;
6. Have donated more than 400 mL of blood within 3 months before screening, or lost more than 400 mL of blood for other reasons, or donated plasma within 14 days before screening;
7. Have used any prescription drugs, vaccines, Chinese herbal medicine within 4 weeks before first dose of the research drug, and/or use any over-the-counter drugs (OTC), vitamins, nutritional supplements within 2 weeks before first dose of the research drug;
8. Have participated in any clinical trial within 3 months before screening;
9. Refuse to stop using any methylxanthine drinks or foods such as coffee, tea, cola, chocolate, or drinks containing grapefruit, or any food that affect the activity of liver enzymes from 48 hours before the first dose of the research drug to the end of the study;
10. Have undergone surgery within 6 months before screening, or plan to receive a surgery recently ;
11. Have abnormality or clinical significance in any infection screening;
12. Have special requirements on diet and cannot accept unified diet;
13. Have the difficulty in venous blood taking or can not tolerate venipuncture, or have a history of dizziness in blood taking;
14. Any other condition that researchers believe unsuitable for enrolling into the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax | Pharmacokinetic plasma samples collected over 36 hour period
  Cmax - Maximum Observed Concentration in Plasma
Bioequivalence based on AUC 0-t | Pharmacokinetic plasma samples collected over 36 hour period
  Area Under the Concentration-time Curve From Time Zero to Time of Last
Bioequivalence based on AUC 0-∞ | Pharmacokinetic plasma samples collected over 36 hour period
  Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institue for Drug Clinical Trials, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No